CLINICAL TRIAL: NCT06266624
Title: Tourniquet-Test in HHT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Freya Droege, Principal Investigator, University Hospital, Essen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Tourniquet in HHT
Record Dates: First submitted 2024-01-12; First posted 2024-02-20 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: HHT
Keywords: HHT; Tourniquet Test
MeSH Terms: interventions — Capillary Fragility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tourniquet Test (Experimental): Patients with HHT patients who undergo the Tourniquet Test
  Interventions: Diagnostic Test: Tourniquet Test

INTERVENTIONS:
Diagnostic Test: Tourniquet Test — Tourniquet Test was performed in patients with HHT

SUMMARY:
The Tourniquet test is used as a diagnostic procedure for thrombocytopathies and vascular diseases. Currently, there is no evidence whether this test is also positive in hereditary haemorrhagic telangiectasia (HHT), a vasculopathy. The aim of this study was to investigate whether this non-invasive test could also be used as an additional diagnostic criterion in patients with HHT.

DETAILED DESCRIPTION:
The Tourniquet test is used as a diagnostic procedure for thrombocytopathies and vascular diseases. Currently, there is no evidence whether this test is also positive in hereditary haemorrhagic telangiectasia (HHT), a vasculopathy. The aim of this study was to investigate whether this non-invasive test could also be used as an additional diagnostic criterion in patients with HHT.

ELIGIBILITY:
Inclusion Criteria:

* In patients with confirmed HHT diagnosis (≥ 3 Curaçao criteria or positive molecular genetics)
* aged over 18 years

Exclusion Criteria:

* if inclusion criteria does not apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
number of positive Tourniquet Test results in HHT patients | three years
  Documentation of the number of positive Tourniquet Test results in HHT patients

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Essen, Essen, Nordrhein Westphalen, Germany

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study are available from the PI on reasonable request.
Supporting Information: Study Protocol